CLINICAL TRIAL: NCT06907342
Title: COSENSE-1: A Feasibility Study for Using a Functional Precision Medicine Platform to Select Oxaliplatin-based Versus Irinotecan-based Chemotherapy Regimens for Patients With Metastatic Colorectal Cancer
Brief Title: Testing a Functional Precision Medicine Approach to Select Chemotherapy for Metastatic Colorectal Cancer (COSENSE-1)
Acronym: COSENSE-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-517677-25-00; 2024-517677-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-21; First posted 2025-04-02 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-03

CONDITIONS: Tumor, Colorectal; Organoids; Tumoroid; Metastatic Colorectal Cancer; Core Needle Biopsy; First-line Treatment
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment cohort (Experimental): FOLFOX or FOLFIRI based on readout from patient-derived tumouroids (via biopsy)
  Interventions: Drug: FOLFOX or FOLFIRI

INTERVENTIONS:
Drug: FOLFOX or FOLFIRI — Treatment allocation from tumouroid readout

SUMMARY:
COSENSE-1 is an unblinded, phase II, single-armed, single center feasibility study for using a functional precision medicine platform to select oxaliplatin-based versus irinotecan-based chemotherapy regimens, for male and female participants aged 18 and older, with microsatellite stable (MSS)/proficient mismatch repair (pMMR) metastatic colorectal cancer (mCRC), that is incurable or not resectable with curative intent.

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to test the feasibility of using a functional precision medicine platform to select oxaliplatin-based versus irinotecan-based chemotherapy regimens for patients with metastatic colorectal cancer. Secondary objectives are to describe the tumour response to treatment using efficacy measures and assess the progression-free survival and the overall survival, and assess the toxicity experienced by the participants. Exploratory objectives include basal research on tumouroids and optimisation of the functional assay to be compatible with clinical practice.

Primary endpoints: The primary endpoints are assessing feasibility:

1. The rate of generating valid tumouroid response reports (valid is defined as a fold-change growth in untreated controls of > 1, registered on day 5, 6, 7 or 8 and normalised with resepect to day 0 or 1): a) per patient included in the trial and b) per patient with successful tumour sample.
2. The time from referral to start of allocated treatment.

Secondary endpoints: Secondary endpoints include efficacy in the form of Response Rates (RR) graded and measured using RECIST v1.1, including Objective Response Rate (ORR), Disease Control Rate (DCR) and Clinical Benefit Rate (CBR), as well as Duration of Response (DoR), Progression Free Survival (PFS), Progression Free Survival Rate at 6 months (PFSR) and Overall Survival (OS). Toxicity will be graded using the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v.5.0).

Trial design and patient population: COSENSE-1 is an unblinded, phase II, single-armed, single-center, consent-based feasibility study for using a functional precision medicine platform to select oxaliplatin-based versus irinotecan-based chemotherapy regimens, for male and female participants aged 18 and older, with microsatellite stable (MSS)/proficient mismatch repair (pMMR) metastatic colorectal cancer (mCRC) that is incurable or not resectable with curative intent. Participants can proceed to the treatment cohort of the trial if standard of care treatment can be allocated within the timeframes given by the Norwegian national recommendations for the treatment of colorectal cancer. The study duration will be up to 36 months for each participant with treatment duration up to 6 months, and the study visit frequency will be one per participant.

Main inclusion criteria:

* ECOG performance status 0 or 1
* Acceptable organ function as defined in Section 5.1 "Inclusion criteria"
* Histologically confirmed pMMR/MSS adenocarcinoma originating from the colon or rectum
* Unresectable metastatic disease (not amenable to radical surgery of the cancer disease at the time of study inclusion)
* The oxaliplatin-based regimen FOLFOX (+/- antibody) versus the irinotecan-based regimen FOLFIRI (+/- antibody), are evaluated by an experienced physician, independent of inclusion in the trial, to be equally recommended for the participant as standard of care first-line therapy in the treatment of mCRC, following the Norwegian national guideline on the treatment of colorectal cancer
* Patient is eligible for full (100%) chemotherapy doses at first treatment cycle

Main exclusion criteria:

* Patient has metastatic MMR deficient/MSI adenocarcinoma
* Patient is ineligible for full (100%) chemotherapy doses at first treatment cycle
* ECOG performance status 2 or worse
* Inability to understand study procedures and comply with them, or disorder that compromises the patient's ability to provide informed consent and/or comply with study procedures
* Patient is not equally eligible for FOLFOX (+/- antibody) and FOLFIRI (+/- antibody) chemotherapy regimens, according to the Norwegian national guideline on the treatment of colorectal cancer

Number of participants:

Approximately 148 patients will be screened to achieve:

1. 133 participants for evaluation of primary and exploratory objectives and endpoints, assessing feasibility.
2. 73 participants for evaluation of all objectives and endpoints, including secondary objectives and endpoints.

Intervention: Oxaliplatin-based or irinotecan-based chemotherapy regimen based on patient-derived tumouroids as guide for clinical decision.

Ethical considerations:

For over two decades, both type of chemotherapy regimens (oxaliplatin-based and irinotecan-based) have been considered equal first-line treatment regimens for this patient group. In clinical practice as of today, no biomarkers are available to guide whether oxaliplatin-based or irinotecan-based chemotherapy will be most effective in treating the individuals' cancer disease. Therefore, treatment typically begins with either regimen, often influenced by local traditions or practices. Furthermore, effectiveness of the chosen regimen is monitored clinically and radiologically, and if efficacy is insufficient or toxicities are intolerable, patients are switched to the alternative regimen after 2-3 months. These months are significant for patients with already limited life expectancy. The COSENSE-1 trial offers a more rational approach by providing the most promising chemotherapy regimen upfront. The prerequisites for COSENSE-1, discards the risk of being allocated to inferior treatment compared to clinical practice, and assures similar time frames, safety and toxicity profiles as in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

General conditions:

1. Age 18 or older
2. ECOG performance status 0 or 1
3. Obtained informed consent
4. Acceptable organ function (defined in publicly available protocol)
5. Women of child-bearing potential and men must agree to use highly effective contraception (defined in publicly available protocol)

   Disease and treatment specific conditions:
6. Histologically confirmed pMMR/MSS adenocarcinoma originating from the colon or rectum
7. Unresectable metastatic disease (not amenable to radical surgery of the cancer disease at the time of study inclusion)
8. Patient has metastatic or primary lesion available for biopsy
9. Patient has measurable or evaluable disease per RECIST (version 1.1)
10. The oxaliplatin-based regimen FOLFOX (+/- antibody) versus the irinotecan-based regimen FOLFIRI (+/- antibody), are evaluated by an experienced physician, independent of inclusion in the trial, to be equally recommended for the participant as standard of care first-line therapy in the treatment of mCRC, following the Norwegian national guideline on the treatment of colorectal cancer (https://www.helsedirektoratet.no/retningslinjer/kreft-i-tykktarm-og-endetarm-handlingsprogram)
11. Patient is eligible for full (100%) chemotherapy doses at first treatment cycle
12. Treatment with chemotherapy can be scheduled within 28 days from referral

Exclusion Criteria:

1. Patient has metastatic MMR deficient/MSI adenocarcinoma
2. Patient is ineligible for full (100%) chemotherapy doses at first treatment cycle
3. Patient is not equally eligible for FOLFOX (+/- antibody) and FOLFIRI (+/- antibody) chemotherapy regimens, according to the Norwegian national guideline on the treatment of colorectal cancer
4. ECOG performance status 2 or worse
5. Pregnancy or planned pregnancy during the study period, due to the risks of drug treatment to a developing foetus
6. Breastfeeding
7. Patients with psychological, geographical, familial or sociological conditions that can prevent compliance with the study protocol
8. Inability to understand study procedures and comply with them, or disorder that compromises the patient's ability to provide informed consent and/or comply with study procedures
9. Patient fulfils any of the contraindications listed in the SmPC of the relevant IMP
10. Treatment cannot be scheduled within 28 days from referral

    Medical history:
11. Partial or complete dihydropyrimidine dehydrogenase (DPD) deficiency
12. Evidence of CNS metastasis
13. Unresolved toxicities of a previous systemic treatment that, in the opinion of the physician, make the patient unfit for inclusion
14. Antitumoural treatment ≤ 30 days before inclusion. Hormonal substitutive treatment is allowed
15. Preexisting significant cardiovascular disease including uncontrolled/unstable or symptomatic angina, uncontrolled atrial or ventricular arrythmias, LVEF known to be < 40% or symptomatic congestive heart failure
16. Stroke (including TIA) or acute myocardial infarction within 6 months before the first dose of study treatment
17. Clinically significant peripheral sensory neuropathy
18. Recent (<6 months before the start of study treatment) pulmonary embolism, deep vein thrombosis, or another significant thromboembolic event
19. History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on chest computed tomography (CT)
20. Evidence of previous acute hypersensitivity reaction to any component of the treatment
21. History of any disease that may increase the risks associated with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2040-09 (Estimated)

PRIMARY OUTCOMES:
Test the feasibility of using a functional precision medicine platform to select oxaliplatin-based versus irinotecan-based chemotherapy regimens for patients with metastatic colorectal cancer. | Up to 1 month
  Rate of generating valid* tumouroid response reports per patient included in the trial. *A valid tumouroid response report for a sample is defined as a fold-change growth in untreated controls of > 1, registered on day 5, 6, 7 or 8 and normalised with respect to day 0 or 1.
Test the feasibility of using a functional precision medicine platform to select oxaliplatin-based versus irinotecan-based chemotherapy regimens for patients with metastatic colorectal cancer. | Up to 1 month
  Rate of generating valid* tumouroid response reports per patient with obtained tumour sample. *A valid tumouroid response report for a sample is defined as a fold-change growth in untreated controls of > 1, registered on day 5, 6, 7 or 8 and normalised with resepect to day 0 or 1.
Test the feasibility of using a functional precision medicine platform to select oxaliplatin-based versus irinotecan-based chemotherapy regimens for patients with metastatic colorectal cancer. | Up to 1 month
  What is the time from referral to start of allocated treatment

SECONDARY OUTCOMES:
Describe the tumour response to treatment using RECIST v.1.1 | Up to 48 months
  Objective Response Rate (ORR)
Describe the tumour response to treatment using RECIST v.1.1 | Up to 48 months
  Disease Control Rate (DCR)
Describe the tumour response to treatment using RECIST v.1.1 | Up to 48 months
  Clinical Benefit Rate (CBR), defined as the percentage of patients who had a complete response, partial response, or had stable disease for 6 months or more
Describe the tumour response to treatment using RECIST v.1.1 | Up to 48 months
  Duration of Response (DoR)
Assess progression free survival | Up to 5 years
  Progression Free Survival (PFS), defined as the time from starting first-line treatment to the time of documentation of progressive disease (PD) according to RECIST v.1.1 on active therapy, determined failure of treatment strategy or death
Assess progression free survival rate | Up to 6 months
  Progression Free Survival Rate (PFSR), defined as the ratio of participants with PFS at 6 months
Assess overall survival | Up to 5 years
  Overall Survival
Toxicity experienced in the trial | Up to 2 years
  Incidence of grade 3-5 adverse events using CTCAE v.5.0

CONTACTS AND LOCATIONS:
Locations (1):
- St. Olavs Hospital, Trondheim, Norway